CLINICAL TRIAL: NCT02943902
Title: An Open-labeled, Randomized Controlled Trial Evaluating for Non-inferiority of 1+1 Compared to 2+1 Dosing Schedules of 10-valent and 13-valent Pneumococcal Conjugate Vaccine (PCV) in South African Children
Brief Title: Reduced PCV Dosing Schedules in South African Infants
Acronym: PCV1+1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Shabir Madhi, Investigator, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCV1+1
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Pneumonia; Meningitis
Keywords: immunogenicity
MeSH Terms: conditions — Pneumonia; Meningitis | interventions — Pneumococcal Vaccines; 10-valent pneumococcal conjugate vaccine; PHiD-CV vaccine; Cornified Envelope Proline-Rich Proteins; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1a (1+1, 6 weeks) (Experimental): PCV10 (Synflorix 0.5ml injection) will be administered at 6 weeks and 9 months of age
  Interventions: Biological: Pneumococcal conjugate vaccine (PCV10 ) 1+1, 6 weeks
- Group 1b (1+1, 6 weeks) (Experimental): PCV13 (Prevenar 13, 0.5ml injection) will be administered at 6 weeks and 9 months of age
  Interventions: Biological: Pneumococcal conjugate vaccine (PCV13 ) 1+1, 6 weeks
- Group 2a (1+1, 14 weeks) (Experimental): PCV10 (Synflorix 0.5ml injection) will be administered at 14 weeks and 9 months of age
  Interventions: Biological: Pneumococcal conjugate vaccine (PCV10 ) 1+1, 14 weeks
- Group 2b (1+1, 14 weeks) (Experimental): PCV13 (Prevenar 13, 0.5ml injection) will be administered at 14 weeks and 9 months of age
  Interventions: Biological: Pneumococcal conjugate vaccine (PCV13 ) 1+1, 14 weeks
- Group 3a (2+1) (Active Comparator): PCV10 (Synflorix 0.5ml injection) will be administered at 6 weeks, 14 weeks and 9 months of age, as per EPI schedule in South Africa
  Interventions: Biological: Pneumococcal conjugate vaccine (PCV10 ) 2+1
- Group 3b (2+1) (Active Comparator): PCV13 (Prevenar 13, 0.5ml injection) will be administered at 6 weeks, 14 weeks and 9 months of age, as per EPI schedule in South Africa
  Interventions: Biological: Pneumococcal conjugate vaccine (PCV13 ) 2+1

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine (PCV10 ) 1+1, 6 weeks — PCV10 1+1, 6 weeks & 9 months
  Other Names: Synflorix (PCV10)
  Arms: Group 1a (1+1, 6 weeks)
Biological: Pneumococcal conjugate vaccine (PCV10 ) 1+1, 14 weeks — PCV10 1+1, 14 weeks & 9 months
  Other Names: Synflorix (PCV10)
  Arms: Group 2a (1+1, 14 weeks)
Biological: Pneumococcal conjugate vaccine (PCV10 ) 2+1 — PCV10 2+1, 6&14 weeks & 9 months
  Other Names: Synflorix (PCV10)
  Arms: Group 3a (2+1)
Biological: Pneumococcal conjugate vaccine (PCV13 ) 1+1, 6 weeks — PCV13 1+1, 6 weeks & 9 months
  Other Names: Prevenar 13
  Arms: Group 1b (1+1, 6 weeks)
Biological: Pneumococcal conjugate vaccine (PCV13 ) 1+1, 14 weeks — PCV13 1+1, 14 weeks & 9 months
  Other Names: Prevenar 13
  Arms: Group 2b (1+1, 14 weeks)
Biological: Pneumococcal conjugate vaccine (PCV13 ) 2+1 — PCV13 2+1, 6&14 weeks & 9 months
  Other Names: Prevenar 13
  Arms: Group 3b (2+1)

SUMMARY:
This study will evaluate the immunogenicity of a reduced dosing schedule of Pneumococcal Conjugate vaccine (PCV) PCV10 and PCV13, in which children will receive a primary dose at either 6 or 14 weeks of age, followed by a booster dose at 9 months of age (1+1 schedule), and compare this immune response to those who receive a two dose primary series (at 6 and 14 weeks of age) and booster dose at 9-months (2+1 schedule).

DETAILED DESCRIPTION:
Pneumonia is the leading global cause of childhood death outside of the neonatal period, and contributes to 19% of the 10 million childhood deaths occurring annually, the majority of which occurs in industrialising countries. Despite the successes in improving primary healthcare in South Africa since 1994, pneumonia nevertheless remains a leading cause of childhood death in South Africa, aggravated by the HIV/AIDS epidemic. Streptococcus pneumoniae is recognised as the leading bacterial cause of pneumonia in children as well as having been identified as a common cause of super-imposed bacterial infection in individuals with respiratory virus-associated pneumonia.

In South Africa, the cost of procurement of PCV ($20 per dose) totals almost 50% of the total cost of all vaccines purchased for the national immunisation program. Similarly, PCV is the most expensive vaccine purchased by the Global Alliance for Vaccines and Immunisation (GAVI), which heavily funds vaccine procurement for low income countries. The sustainability of continued procurement of this vaccine at the current pricing in low-middle income countries remains uncertain.

This will be a randomized, open-label study (laboratory personnel will however be blinded) in which subjects are randomized to one of two (primary dose at either 6 or 14 weeks of age) 1+1 dosing schedules of PCV10 or PCV13, or to a 2+1 schedule of these vaccines. A total of 600 subjects will be randomized in a 1:1:1:1:1:1 ratio to one of the six groups. The study will be undertaken at an experienced research site in Johannesburg, South Africa, where the 600 children born to HIV-uninfected women are expected to be enrolled over a 12- month period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the parent/guardian of the child;
2. Born to an HIV-uninfected women, based on testing undertaken as part of standard of care during the last trimester of pregnancy;
3. Had not received any vaccine other than BCG and OPV (routinely given at birth) prior to enrolment;
4. Birth weight >2499g AND weight of child >3.5 kg at time of proposed randomization;
5. Aged 42-56 days of age at time of enrolment;
6. Available for the duration of the study;
7. Child is healthy based on medical history and physical examination of the study-staff.

Exclusion Criteria:

1. Any clinically significant major congenital abnormalities;
2. Previous hospitalization for a respiratory illness following discharge from hospital after birth;
3. Receipt of any other investigational drug/vaccine. Co-enrollment into non-investigational studies, including epidemiology studies, is allowed;
4. Any previous PCV vaccination;
5. Known allergy to any of the vaccine components;
6. Febrile illness (axillary temperature ≥37.8°C) at time of enrolment. These participants are eligible if the temperature resolves for at least 48 hours and they remain within the study defined window periods;
7. Planned relocation to outside of the study area during up until age of 2 years;
8. Receipt of blood transfusion or any other blood products (including immunoglobulins) since birth. Receipt of such products during the course of the study, will require withdrawal of the child from the study;
9. History of confirmed pneumococcal disease since birth;
10. Any known or suspected immunodeficiency condition which could affect immune response to vaccination.

Ages: 5 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
serotype specific geometric mean antibody concentrations (GMC) one month following the booster dose | 1 month post booster vaccine
  The serotype-specific GMC measured 1 month after the 9-month booster dose for each 1+1 vaccine group and comparing it to the 2+1 group of the same vaccine

SECONDARY OUTCOMES:
Immunogenicity: percentage of children with vaccine-serotype specific serum IgG antibody concentration above the WHO-defined putative threshold for protection (≥0.35 µg/mL) at 9 months of age, prior to the booster dose of differing 1+1 dosing schedules | 9 months of age
  1. To evaluate the percentage of children with vaccine-serotype specific serum IgG antibody concentration above the WHO-defined putative threshold for protection (≥0.35 µg/mL) at 9 months of age, prior to the booster dose of differing 1+1 dosing schedules (i.e. primary dose given at either 6 or 14 weeks of age) compared to that of children who received a 2 dose primary series (i.e. 2+1 dosing schedule group)..

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MD, PhD, Principal Investigator — University of Witwatersrand, South Africa
Locations (2):
- South Africa (2):
  - Chris Hani Baragwanath Academic Hospital, Johannesburg, Gauteng
  - Nrf/Dst Vpd Rmpru, Soweto, GP

IPD SHARING:
Plan to Share IPD: Yes
The data will be made publically available, within one year of completion of the study to any investigators or BMGF nominated partners, who wish to use the data to address any specific questions not directly addressed under the study objectives and which the data would lend itself to

REFERENCES:
- [Derived] Izu A, Mutsaerts EA, Olwagen C, Jose L, Koen A, Nana AJ, Cutland CL, Madhi SA. Serotype-specific serum immunoglobulin G at 18 months of age following one or two doses of a primary series of 10-valent or 13-valent pneumococcal conjugate vaccine and a booster dose at nine months of age: a randomized controlled study. Expert Rev Vaccines. 2025 Dec;24(1):121-127. doi: 10.1080/14760584.2025.2458179. Epub 2025 Jan 27. PMID 39865559
- [Derived] Mutsaerts EAML, van Cranenbroek B, Madhi SA, Simonetti E, Arns AJ, Jose L, Koen A, van Herwaarden AE, de Jonge MI, Verhagen LM. Impact of nutritional status on vaccine-induced immunity in children living in South Africa: Investigating the B-cell repertoire and metabolic hormones. Vaccine. 2024 May 22;42(14):3337-3345. doi: 10.1016/j.vaccine.2024.04.034. Epub 2024 Apr 17. PMID 38637212
- [Derived] Olwagen CP, Izu A, Mutsaerts EAML, Jose L, Koen A, Downs SL, Van Der Merwe L, Laubscher M, Nana AJ, Moultrie A, Cutland CL, Dorfman JR, Madhi SA. Single priming and booster dose of ten-valent and 13-valent pneumococcal conjugate vaccines and Streptococcus pneumoniae colonisation in children in South Africa: a single-centre, open-label, randomised trial. Lancet Child Adolesc Health. 2023 May;7(5):326-335. doi: 10.1016/S2352-4642(23)00025-1. Epub 2023 Mar 16. PMID 36934731
- [Derived] Madhi SA, Mutsaerts EA, Izu A, Boyce W, Bhikha S, Ikulinda BT, Jose L, Koen A, Nana AJ, Moultrie A, Roalfe L, Hunt A, Goldblatt D, Cutland CL, Dorfman JR. Immunogenicity of a single-dose compared with a two-dose primary series followed by a booster dose of ten-valent or 13-valent pneumococcal conjugate vaccine in South African children: an open-label, randomised, non-inferiority trial. Lancet Infect Dis. 2020 Dec;20(12):1426-1436. doi: 10.1016/S1473-3099(20)30289-9. Epub 2020 Aug 25. PMID 32857992